CLINICAL TRIAL: NCT00143689
Title: A Pilot Study of a Nucleoside Analogue Reverse Transcriptase Inhibitor Sparing Regimen in Antiretroviral-Naïve, HIV-infected Patients
Brief Title: NRTI-Sparing Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Abbott (Industry); Boehringer Ingelheim (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H02-50066; CTN 177
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV; Mitochondrial Toxicity
MeSH Terms: interventions — Lopinavir; Ritonavir; Nevirapine; Zidovudine; Lamivudine

ARMS (1):
- Lopinavir/ritonavir, Zidovudine, Lamivudine (Experimental): Participants will be randomly assigned to receive one of the following drug combinations:
  * lopinavir/ritonavir (Kaletra) and nevirapine (Viramune) twice a day;
  * Combivir (Zidovudine (AZT) plus lamivudine (3TC)) and nevirapine twice a day;
  * Combivir and lopinavir/ritonavir twice a day.
  Interventions: Drug: lopinavir/ritonavir; nevirapine; Zidovudine; Lamivudine

INTERVENTIONS:
Drug: lopinavir/ritonavir; nevirapine; Zidovudine; Lamivudine — See Detailed Description.

SUMMARY:
This study will compare a nucleoside reverse transcriptase inhibitor-sparing (NRTI-sparing) regimen (Kaletra + nevirapine) to two nucleoside reverse transcriptase inhibitor-based regimens (Combivir + nevirapine and Combivir + Kaletra).

Participants will be randomly assigned to receive one of the following drug combinations:

* lopinavir/ritonavir (Kaletra) and nevirapine (Viramune) twice a day;
* Combivir (Zidovudine (AZT) plus lamivudine (3TC)) and nevirapine twice a day;
* Combivir and lopinavir/ritonavir twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Be HIV-positive
* Be at least18 years of age
* Have viral load above 5 000 copies/ml
* Be likely to comply with the study protocol
* Agree not to take, for the duration of the study, any drug that is contraindicated with the study drugs
* Agree not to take any medication, including over-the-counter medicine, alcohol, or street drugs without the knowledge and permission of the principal investigator

Exclusion Criteria:

* Have ever received antiretroviral therapy
* Pregnancy or breastfeeding
* Have abnormal laboratory tests (see investigator)
* Have received an investigational drug within 30 days of study drugs administration
* Be receiving systemic chemotherapy
* Have an acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Changes in mitochondrial DNA/Nuclear DNA (mtDNA/nDNA) ratio at 48 weeks, as a marker of mitochondrial toxicity. | 48 weeks

SECONDARY OUTCOMES:
Changes in mitochondrial DNA/Nuclear DNA (mtDNA/nDNA) ratio at 96 weeks | 96 weeks
Proportions of patients with viral load below 50 and below 400 copies/mL
Viral load changes from baseline
Rates and extent of immune reconstitution (CD4 count increase)
Rates and severity of dyslipidemia and insuline resistance/diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Julio Montaner, MD, Principal Investigator — University of British Columbia/Providence Health Care
Locations (4):
- Canada (4):
  - McMaster University, Hamilton, Ontario
  - University of Ottawa Health Services, Ottawa, Ontario
  - Maple Leaf Clinic, Toronto, Ontario
  - Clinique Medicale L'Actuel, Montreal, Quebec